CLINICAL TRIAL: NCT03172169
Title: Observational Study of Specific Small RNA in Plasma Muscle Tissue for Predicting Diaphragm Dysfunction in Mechanically Ventilated Patients
Brief Title: Specific Small RNA in Plasma for Predicting Diaphragm Dysfunction in Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Principal Investigator, Southeast University, China
Other Study IDs: miRNA and Diaphragm
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group: no intervention
  Interventions: Other: no Intervention
- Difficult withdrawal group: The mechanical ventilation time was >48 hours and the first SBT failure
  Interventions: Other: no Intervention
- Mechanical ventilation control group: Elective and expected postoperative control of mechanical ventilation time greater than 12h after cardiothoracic surgery
  Interventions: Other: no Intervention

INTERVENTIONS:
Other: no Intervention — no Intervention

SUMMARY:
Through the literature screening of MyomiRX 7, the detection of mechanical ventilation group, difficult withdrawal unit and healthy adult plasma levels of MyomiRX in the evaluation of function and skeletal muscle thickness of the diaphragm, the correlation analysis of 7 kinds of MyomiRX and diaphragmatic dysfunction. The research value of this project is to explore the predictive value of plasma MyomiRX level on diaphragmatic dysfunction in patients with mechanical ventilation, and to lay the foundation for finding the target of VIDD diagnosis and treatment

DETAILED DESCRIPTION:
1. research content (1) screening MyomiR through literature review (2) selection of mechanical ventilation group, difficult withdrawal units and three healthy adult groups, method for the detection of plasma MyomiRX level and clinical assessment of diaphragmatic function, observation of the relationship between MyomiRX level and diaphragmatic dysfunction, prediction of plasma MyomiRX levels in patients with mechanical ventilation for diaphragmatic dysfunction in value.
2. research objectives Objective to investigate the predictive value of specific minute RNA in plasma muscle tissue on diaphragmatic dysfunction in mechanical ventilation patients Experimental grouping (1) the control group of mechanical ventilation (time of examination, preoperative, admission to ICU and before extubation); (2) difficulty in withdrawal of units (first days, third days and seventh days after the failure of the test time for the first withdrawal); (3) the healthy control group (after the test time was selected)

ELIGIBILITY:
Inclusion Criteria:

healthy control group: healthy volunteers mechanical ventilation control group: patients who underwent elective cardiothoracic surgery after scheduled and controlled mechanical ventilation for more than 12h were transferred to ICU (including coronary artery bypass grafting and valve replacement) difficult weaning: difficult to diagnose patients in ICU (weaning time from mechanical ventilation for >48 hours and first SBT failure)

Exclusion Criteria:

1. severe respiratory depression, high paraplegia and neuromuscular lesions;
2. esophageal obstruction, esophageal perforation, severe esophageal varices bleeding, upper gastrointestinal surgery and other reasons can not be placed EAdi catheter;
3. thoracic deformity and diaphragmatic hernia;
4. serious heart, liver, kidney and other organ failure, hemodynamic instability;
5. pregnancy;
6. the end of the tumor or the family member give up the active treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy control group: healthy volunteers mechanical ventilation control group: patients who underwent elective cardiothoracic surgery after scheduled and controlled mechanical ventilation for more than 12h were transferred to ICU (including coronary artery bypass grafting and valve replacement) difficult weaning: difficult to diagnose patients in ICU (weaning time from mechanical ventilation for >48 hours and first SBT failure)
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of diaphragmatic dysfunction using RT-PCR microRNA level | 7 days
  Prediction of diaphragmatic dysfunction in patients with mechanical ventilation by specific minute RNA of plasma muscle tissue

CONTACTS AND LOCATIONS:
Overall Officials: pan chun, doctor, Principal Investigator — Colleague

IPD SHARING:
Plan to Share IPD: Undecided